CLINICAL TRIAL: NCT07210515
Title: A Randomized, Triple-blind, Placebo-controlled, Phase 3 Trial to Evaluate the Efficacy, Safety, and Tolerability of Intravenous AMBTX-01 (Neridronate) for Treatment of Complex Regional Pain Syndrome Type 1 (CRPS-RISE)
Brief Title: Evaluation of IV AMBTX-01 (Neridronate) for Treatment of CRPS Type 1 (CRPS-RISE)
Acronym: CRPS-RISE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ambros Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMBTX-01-301
Record Dates: First submitted 2025-09-17; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Complex Regional Pain Syndrome Type I
Keywords: CRPS; edema; pain; RDS
MeSH Terms: conditions — Complex Regional Pain Syndromes; Edema; Pain | interventions — 6-amino-1-hydroxyhexane-1,1-diphosphonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- neridronate (Experimental): 400 mg AMBTX-01 infusion
  Interventions: Drug: Neridronate
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neridronate — neridronate 100 mg, given as a 2-hour infusion on Days 1, 4, 7, and 10.
  Arms: neridronate
Drug: Placebo — placebo comparator
  Arms: Placebo

SUMMARY:
Phase 3 Trial of AMBTX-01 (neridronate) for Complex Regional Pain Syndrome Type 1

DETAILED DESCRIPTION:
This is a multicenter, randomized, triple-blind, controlled trial, to assess the efficacy, safety, and tolerability of neridronate 400 mg IV in adult participants with the warm subtype of Complex Regional Pain Syndrome Type 1 (CRPS-1) and a positive triple phase bone scan (TPBS).

The total planned trial duration for each participant will be approximately up to 18 weeks and will include:

* Screening period of up to 6 weeks
* Treatment period on Days 1, 4, 7, and 10
* Post-treatment follow-up through week 12

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant ≥ 18 years of age at time of Screening.
2. A diagnosis of CRPS-1 according to the clinical Budapest Criteria as recommended by the International Association for the Study of Pain (IASP), as well as no known peripheral nerve injury. Signs and symptoms of CRPS must apply to a single identified affected limb (i.e., arm, hand, wrist, leg, ankle or foot) and must demonstrate asymmetry with respect to the contralateral limb.
3. Single affected limb at the Screening and Randomization Visits meeting the following warm subtype criteria:

   1. Edema in the affected limb
   2. AND ≥ 2 of the following:

      1. Obvious redness in the affected region relative to the same region on the contralateral limb on inspection
      2. ≥ 1°C increase in temperature on the affected limb relative to the contralateral limb
      3. Moderate-to-severe edema
4. CRPS symptoms ≤ 6 months since onset.
5. Increased uptake in the involved limb compared to the contralateral limb on TPBS (phase 2 and/or phase 3) during Screening. A historic scan not older than 3 months prior to Randomization Visit is acceptable, if available and of sufficient quality for a central read.
6. "Pain now" assessments of > 4 on the 11 point numerical rating scale in the CRPS affected limb.
7. Women of childbearing potential must:

   1. Be nonpregnant.
   2. Be nonlactating.
   3. Agree to use a highly effective method of contraception and for at least 6 months following last investigational product administration.

Exception: Women exclusively engaging in same sex sexual activities are not required to meet this criterion.

Exclusion Criteria

1. A current or prior diagnosis of CRPS Type 2 or CRPS not otherwise specified (CRPS NOS), or whose CRPS has no known inciting event, or CRPS-1 without criteria of the warm subtype at the time of Screening.
2. ≥ 40 points on the Pain Catastrophizing Scale.
3. Prior use of neridronate or participation in a clinical study where the participant may have received neridronate.
4. Participants currently taking or planning to be treated with prohibited concomitant medications/therapies, or not likely able to follow the protocol restrictions for use of concomitant treatment.
5. Severely impaired renal function.
6. Hypocalcemia.
7. Vitamin D deficiency.
8. Significant dental findings such as an unhealed tooth extraction site.
9. Eye inflammation.
10. Significantly elevated liver-related lab tests or evidence of significant liver disease.
11. Clinically unstable cardiac disease.
12. Any known conditions, from 3 months prior to Screening Visit or to the Randomization Visit, that may interfere with the assessment of CRPS-1, CRPS-related pain, safety, or other trial assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to Week 12. | Week 12
  Assessed on an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 representing the worst possible pain.

SECONDARY OUTCOMES:
At least a 50% reduction from baseline to Week 12 in pain intensity. | Week 12
  Assessed using an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain.
Change from baseline in CRPS Severity Score (CSS) to Week 12. | Week 12
  Assessed using the CRPS CSS, a 0-16 scale where higher scores denotes greater CRPS symptom severity and lower scores reflect milder symptoms.
Patient Global Impression of Change (PGI-C) in CRPS-Related Health. | Week 12
  Assessed using the PGI-C, a 7-point numerical rating scale where 1 indicates "very much improved" and 7 indicates "very much worse."
Change from baseline in the Short Form 36 (SF-36) Item Health Survey Physical Functioning domain. | Week 12
  Assessed using the SF-36, a validated 36-item self-reported questionnaire that measures health-related quality of life across eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores range from 0 to 100, with higher scores indicating better health status.
Change from baseline over time in pain intensity. | Day 10, Weeks 3, 6, and 9
  Assessed on an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 representing the worst possible pain.
At least a 50% reduction from baseline in pain intensity. | Days 10, Weeks 3, 6, and 9
  Assessed using an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain.
At least a 30%, 70%, and 90% reduction from baseline in pain intensity. | Day 10, Weeks 3, 6, 9, and 12
  Assessed using an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain.
Time to onset of analgesic improvement. | daily assessment up to week 12
  Assessed as the time to onset of analgesic improvement, defined by a ≥30% reduction in pain intensity from baseline, based on the 7-day average of twice-daily "pain now" ratings on the 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain. The improvement must be sustained for a minimum of one week.
Time to at least a 50%, 70%, and 90% reduction from baseline in pain intensity. | 7-day average
  Assessed using an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain.
Change from baseline in the 7-day average of the twice-daily "worst possible pain" assessments. | 7-day average
  Assessed using the average score from the 11-point Numerical Rating Scale (NRS), where 0 denotes no pain and 10 denotes the worst possible pain
At least a 30%, 50%, 70%, and 90% reduction from baseline in pain intensity. | Day 10, Weeks 3, 6, 9, and 12
  Assessed using an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain.
Change from baseline in pain evoked by active motion. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed using an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain in the CRPS affected limb.
At least a 50% reduction from baseline in pain evoked by active motion. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed using an 11-point Numerical Rating Scale (NRS), with 0 representing no pain and 10 the worst possible pain in the affected limb.
Change from baseline in active range of motion (AROM) of affected limb vs. contralateral limb. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed by measuring range of motion of selected joints using a goniometer, and calculating the change from baseline for each joint assessed.
Change from baseline in the CRPS Severity Score (CSS) and in the individual elements of the CRPS Severity Score. | Days 4, 7, 10, Weeks 3, 6, and 9
  CRPS severity score is a series of 17, 0-1 questions (where 0 is that the sign/symptom is not displayed and 1 is that the sign/symptom is displayed) and scored for a total score of 0 (no CRPS signs/symptoms) to 17 (worse CRPS severity).
Change from baseline in edema of affected limb. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed using the "edema" using 4-point numerical rating scale where 0 is no edema and 3 is severe edema.
Change from baseline in temperature of affected limb vs contralateral limb. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessment of 'temperature' is defined as the difference in temperature, measured in degrees Celsius (°C) using an infrared thermometer, between the affected limb and the contralateral limb.
Change from baseline in use of rescue analgesic medications. | Day 10, Weeks 3, 6, 9, and 12
  Changes from baseline at each time point will be classified as improved (yes-to-no), unchanged (no-to-no or yes-to-yes), or worsened (no-to-yes).
Change from baseline in mean daily dose of rescue analgesic medicines. | Day 10, Weeks 3, 6, 9, and 12
  Assessed as the mean daily dose of rescue analgesic medications, calculated over the 7-day period preceding each scheduled timepoint.
Change from baseline in heavy use of rescue analgesic medications. | Day 10, Weeks 3, 6, 9, and 12
  Changes from baseline at each time point will be classified as improved (yes-to-no), unchanged (no-to-no or yes-to-yes), or worsened (no-to-yes) where "heavy use" is defined as ≥ 3000 mg acetaminophen > 3 days/week and/or ≥ 15 mg oxycodone > 3 days/week during the 7 days before the given study visit.
Patient Global Impression of Change (PGI-C) in CRPS-related health. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed using a categorical scale of: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," and "very much worse," which will be mapped to numeric values of -3, -2, -1, 0, 1, 2, and 3, respectively.
Clinician Global Impression of Change (CGI-C) in CRPS-related health. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed using a categorical scale of: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," and "very much worse," which correspond to numeric values of 0, 1, 2, 3, 4, and 5, respectively.
Change from baseline in Patient Global Impression of Severity (PGI-S) in CRPS Severity. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed using a categorical scale of: "none," "minimal," "mild," "moderate," "severe," and "very severe," which will be mapped to numeric values of -3, -2, -1, 0, 1, 2, and 3, respectively.
Change from baseline in Short Form McGill Pain Questionnaire (SF-MPQ) (a) Total Pain Score, (b) each of 4 domain scores, (c) single items. | Days 4, 7, 10, and Weeks 3, 6, 9, and 12
  Assessed using a response to 22 descriptors rated on an 11-point numerical scale (NRS), capturing both neuropathic and non-neuropathic aspects. These descriptors are grouped into four core domains-Continuous Pain, Intermittent Pain, Neuropathic Pain, and Affective Descriptors-with domain scores calculated as the mean of items within each domain. The overall pain score is derived from the average of the 22 items. The complete scale runs from 0 to 10, where a higher score represents greater pain severity.
Moderate (at least 30%) and substantial (at least 50%) improvement in Short Form McGill Pain Questionnaire (SF-MPQ) (a) Total Pain Score, and (b) each of 4 domain scores. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessed using a response to 22 descriptors rated on an 11-point numerical scale (NRS), capturing both neuropathic and non-neuropathic aspects. These descriptors are grouped into four core domains-Continuous Pain, Intermittent Pain, Neuropathic Pain, and Affective Descriptors-with domain scores calculated as the mean of items within each domain. The overall pain score is derived from the average of the 22 items. The complete scale runs from 0 to 10, where a higher score represents greater pain severity.
Change from baseline in the Short Form 36 (SF-36) Item Health Survey (a) 8 domain scores and (b) 2 component summary scores. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessment focuses on changes across eight domains: Physical Functioning, Role Limitations due to Physical Health, Role Limitations due to Emotional Problems, Energy/Fatigue, Emotional Well-being, and Social Functioning. Two summary scores-Physical Component Summary and Mental Component Summary-are derived. All domain scores are standardized to a 0-100 scale, with higher scores reflecting better health status
Moderate (≥ 30%) and substantial (≥ 50%) improvement in the Short Form 36 (SF-36) Item Health Survey (a) 8 domain scores and (b) 2 component summary scores. | Days 4, 7, 10, Weeks 3, 6, 9, and 12
  Assessment focuses on changes across eight domains: Physical Functioning, Role Limitations due to Physical Health, Role Limitations due to Emotional Problems, Energy/Fatigue, Emotional Well-being, and Social Functioning. Two summary scores-Physical Component Summary and Mental Component Summary-are derived. All domain scores are standardized to a 0-100 scale, with higher scores reflecting better health status
Change from baseline in the daily sleep interference scale (DSIS). | Day 10, Weeks 3, 6, 9, and 12
  Assessed using the 7-day average score on the 11-point Numerical Rating Scale (NRS), where 0 represents did not interfere with sleep and 10 represents completely interfered with sleep - unable to sleep due to CRPS pain.
Moderate (≥ 30%) and substantial (≥ 50%) improvement in the daily sleep interference scale (DSIS). | Day 10, Weeks 3, 6, 9, and 12
  Assessed using the 7-day average score on the 11-point Numerical Rating Scale (NRS), where 0 represents did not interfere with sleep and 10 represents completely interfered with sleep - unable to sleep due to CRPS pain.
Time to moderate (≥ 30%) and substantial (≥ 50%) reduction from baseline in the daily sleep interference scale (DSIS). | 7-day average
  Assessed using the 7-day average score on the 11-point Numerical Rating Scale (NRS), where 0 represents did not interfere with sleep and 10 represents completely interfered with sleep - unable to sleep due to CRPS pain.

IPD SHARING:
Plan to Share IPD: Undecided